CLINICAL TRIAL: NCT01282892
Title: Visceral Abdominal Fat, Non Alcoholic Fatty Liver Diseases and Asymptomatic Coronary Atherosclerosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Liver Clinic, Ziv medical center
Other Study IDs: 0052-08
Record Dates: First submitted 2011-01-18; First posted 2011-01-25 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Visceral Fat; Fatty Liver; Atherosclerosis; Coronary Computed Tomography Angiography
Keywords: Visceral fat; fatty liver; atherosclerosis; coronary computed tomography angiography
MeSH Terms: conditions — Fatty Liver; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with NAFLD
  Interventions: Procedure: patients with NAFLD
- excess of visceral fat
  Interventions: Procedure: excess of visceral fat

INTERVENTIONS:
Procedure: excess of visceral fat — excess of visceral fat
  Groups: excess of visceral fat
Procedure: patients with NAFLD — patients with NAFLD
  Groups: patients with NAFLD

SUMMARY:
Visceral fat or peri-omental fat is increasingly associated with metabolic syndrome, a condition carrying a high risk of coronary artery disease. The independent role of Visceral Fat in cardiovascular risk remains unclear.

Patients with excess of visceral fat and NAFLD patients will have higher prevalence of coronary atherosclerosis plaques independently by metabolic syndrome diagnosis. Suggesting that the presence of visceral fat and/or fatty liver will be considered an important condition to optimize the cardiovascular risk stratification

DETAILED DESCRIPTION:
Abstract Background: Visceral fat or peri-omental fat is increasingly associated with metabolic syndrome, a condition carrying a high risk of coronary artery disease. The independent role of Visceral Fat in cardiovascular risk remains unclear. Aim: Evaluate the relationship between visceral fat, fatty liver and asymptomatic coronary atherosclerosis in patients with the major cardiovascular risk factors and with or without metabolic syndrome.

Methods: 50 patients (age 53±7) with excess of visceral fat visceral, 30 patients with NAFLD and 30 sex, age matched individuals without NAFLD will be recruited . All will be asymptomatic for cardiac related symptoms. Subjects with clinical history of ischemic heart disease, cerebrovascular disease, renal failure, cancer and allergy to lode will be excluded. Coronary artery disease (CAD) will be defined as coronary plaques, with obstructive (70%) or non obstructive lesions (30%). Degree of fatty infiltration (ultrasound), Visceral fat amount (CT), coronary plaques and stenosis (coronary computed tomography angiography,CCTA), markers of insulin resistance,lipotoxicity, systemic inflammation, and oxidant-antioxidant status will be measured measured.

Expected Results: Patients with excess of visceral fat and patients with NAFLD will have higher prevalence of coronary plaques and higher prevalence of non obstructive coronary stenosis, higher HOMA CRP, and TG serum levels than controls. In patients with excess of visceral fat , more segments with atherosclerosis per patient will be detected . Multiple regression analysis is expected to show that visceral fat and fatty liver are strong predictors of coronary atherosclerosis independently by metabolic syndrome diagnosis and independently by markers of insulin resistance, lipotoxicity and inflammation.

Conclusion: Patients with excess of visceral fat and NAFLD patients will have higher prevalence of coronary atherosclerosis plaques independently by metabolic syndrome diagnosis. Suggesting that the presence of visceral fat and/or fatty liver will be considered an important condition to optimize the cardiovascular risk stratification.

ELIGIBILITY:
Inclusion Criteria:

* excess of visceral fat with the major cardiovascular risk factors for coronary CT,
* diagnosis of fatty liver defined by the presence of bright liver echo pattern, absence of alcohol use (<20g/day),
* negative serology for hepatitis B or C diagnosis,
* negative auto antibodies,
* absence of history of another known liver disease,
* 30 sex-age-matched individual with cardiovascular risk factors and without NAFLD and without visceral fat will be considered as controls.
* Informed consent will be obtained from each individual and the study will be presented to the the local ethics committee.

Exclusion Criteria:

* subjects with severe obesity (BMI>35),
* recent history of acute illness,
* clinical history of ischemic heart disease and cerebro vascular disease,
* typical chest pain,
* previous coronary artery disease,
* conventional coronary angiography,
* percutaneous interventions,
* coronary by pass grafting,
* renal failure,
* cancer patients,
* subjects who take drugs that induces hepatic steatosis ( corticosteroids, estrogens, methotrexate, amiodarone and others).
* Exclusion criteria for coronary computed tomography angiography will included also the presence of multiple ectopic beats, atrial fibrillation, heart rate more than 75/min despite therapy, severe lung disease, or a history of allergic reaction to iodine-containing contrast agents.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 patients (age 53±7) with excess of visceral fat visceral, 30 patients with NAFLD and 30 sex, age matched individuals without NAFLD will be recruited
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Liver clinic, Safed
  - Ziv medical center liver unit, Safed, Israel